CLINICAL TRIAL: NCT04311749
Title: The Role of Expanded Panel Non-Invasive Prenatal Testing in Identifying Rare Autosomal Trisomies in Pregnancies With Placentally-Mediated Complications
Brief Title: Expanded NIPT for Pregnancy Complications
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 19-27769
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Fetal Growth Restriction; Preeclampsia Severe
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal blood
  * Placental biopsies
  * Umbilical cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fetal growth restriction
  Interventions: Genetic: Expanded panel cell free DNA testing (non-invasive prenatal testing); Genetic: Placental biopsy; Genetic: Umbilical cord blood

INTERVENTIONS:
Genetic: Expanded panel cell free DNA testing (non-invasive prenatal testing) — Maternal blood sampling
Genetic: Placental biopsy — Post-delivery placental sampling
Genetic: Umbilical cord blood — Post-delivery umbilical cord blood sampling

SUMMARY:
This study evaluates the utility of expanded panel non-invasive prenatal testing (NIPT) in detecting confined placental mosaicism of rare autosomal trisomies among pregnancies with placentally-mediated complications, including fetal growth restriction and severe preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early onset (< 34 weeks) severe fetal growth restriction, defined as estimated fetal weight less than 10th percentile with abnormal umbilical artery Dopplers OR estimated fetal weight less than 5th percentile alone OR biometric size at least 14 days behind expected dates

Exclusion Criteria:

* Maternal age < 18 years
* Multifetal gestation
* Chronic hypertension require use of pharmacotherapy
* Tobacco or drug use
* Major congenital malformations

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: This study includes pregnant women diagnosed with severe, early onset, unexplained fetal growth restriction.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Composite adverse pregnancy outcome | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Preterm birth < 34 weeks | Through study completion, an average of 2 years
Neonatal intensive care unit admission | Through study completion, an average of 2 years
Intrauterine fetal demise | Through study completion, an average of 2 years
  Death of fetus prior to delivery
Neonatal demise | Through study completion, an average of 2 years
  Death of infant within 28 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Sobhani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No